CLINICAL TRIAL: NCT07030725
Title: Targeted TRPM8 Stimulation and Brown Adipose Tissue Activation in Humans
Brief Title: Menthol Stimulation of Brown Adipose Tissue in Humans: Aim 1
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Blair D. Johnson, PhD, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 24695
Record Dates: First submitted 2025-03-07; First posted 2025-06-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Regulation of Energy Expenditure
Keywords: menthol; brown adipose tissue; energy expenditure
MeSH Terms: interventions — salicylhydroxamic acid; Flowering time control protein FCA, Arabidopsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Menthol (Experimental): Menthol (5% L-menthol) applied to the anterior upper body, excluding the arms, head, and neck.
  Interventions: Drug: Menthol Gel
- Sham (Sham Comparator): A sham cream applied to the anterior upper body, excluding the arms, head, and neck.
  Interventions: Drug: Sham
- Time control (Other): No cream applied to the anterior upper body.
  Interventions: Behavioral: Time control

INTERVENTIONS:
Drug: Menthol Gel — Menthol (5% L-menthol) will be applied to the anterior thorax.
  Arms: Menthol
Drug: Sham — Sham gel applied to the anterior thorax.
  Arms: Sham
Behavioral: Time control — No gel applied to anterior thorax.
  Arms: Time control

SUMMARY:
Brown adipose tissue becomes activated during cold conditions to increase thermogenesis (i.e., energy expenditure). Topical menthol application increases resting energy expenditure but it is unclear whether brown adipose tissue activation contributes to this rise in the energy expenditure. The overall goal with this project is to determine whether topical menthol application stimulates brown adipose tissue.

DETAILED DESCRIPTION:
Brown adipose tissue (BAT) is an important organ in the regulation of energy balance, particularly in small mammals and infants. Until recently, BAT was thought to be nonexistent and thus metabolically irrelevant in adult humans, primarily due to the lack of methods capable of localizing and measuring its metabolic contribution. Since its discovery in adult humans, various reports have shown that BAT can be activated in response to cold exposure to increase non-shivering thermogenesis (NST). NST results primarily from the expression of uncoupling protein 1 (UCP1) in BAT, dissipating the energy of the proton motive force as heat, thus uncoupling it from mitochondrial respiration. Notably, activation of BAT augments glucose uptake, improving glucose regulation and insulin sensitivity. Whereas mild cold exposure and beta-3-adrenergic pharmacological stimulation have previously been used to augment BAT-induced thermogenesis, recent investigations have proposed novel methods for UCP1 expression.

Menthol, a chemical cooling agent naturally produced from mint oils, elicits a cold sensation when topically applied to the skin and is used clinically as a pain analgesic. This sensation is derived from the activation of cold-sensitive receptors known as transient receptor potential melastatin 8 (TRPM8), a primary sensor of thermal stimuli in the peripheral nervous system. While TRPM8 is predominately located on the cell membrane of sensory neurons, its expression has been recently detected on BAT, highlighting a potential alternative avenue for stimulating this highly thermogenic tissue. Previous reports have alluded to menthol's potential as a vehicle for BAT activation. Vizin et. al observed a persistent increase in energy expenditure following a short-term topical menthol intervention in a rodent model. Moreover, Valente et. al observed an increase in metabolic rate in humans following a single administration of menthol to the skin surface of the neck and of the right arm and leg. While both groups attribute their findings to menthol-induced BAT activation, there were no markers of BAT activation utilized in their investigations. Therefore, there is a significant scientific gap in the understanding of menthol-induced thermogenesis.

Despite the promising thermogenic potential of topical menthol application, the previously reported increase in metabolic rate may be attributed to other forms of thermogenesis, such as shivering thermogenesis and NST in skeletal muscle. Furthermore, methodological differences regarding application site/area, dosage of menthol, evaporative potential of the skin, and resting vasomotor tone complicate most studies in this field, providing limited clarity on the link between TRPM8 stimulation and UCP1-dependent NST. Due to this, proper characterization of menthol's influence, specifically on physiological responses that contribute to human thermoregulation, is warranted.

Specific Aim: Determine the specific thermogenic mechanism(s) underlying the increase in energy expenditure evoked by menthol induced TRPM8 activation.

Hypothesis: Topical menthol application to the anterior aspect of the thorax will increase thermogenesis (i.e., resting energy expenditure) via activation of BAT (i.e., supraclavicular skin temperature; indirect-noninvasive measure of BAT activity) and augmentation of skeletal muscle blood flow (i.e., estimated via changes in limb blood flow) versus application of a sham cream.

ELIGIBILITY:
Inclusion Criteria:

* Fluency in English
* Participate in 150 minutes or more of at least moderate intensity exercise per week during the previous year. Assessment of moderate intensity physical activity will be determined via the International Physical Activity Questionnaire (i.e., IPAQ) (described in detail in Section 7.0). This questionnaire defines moderate intensity exercise as "activities that take moderate physical effort and make you breathe somewhat harder than normal".
* Body fat ≤ 30% as determined by DEXA scan
* Be cleared for physical activity according to the 2020 Physical Activity Readiness Questionnnaire (PAR-Q+).

Exclusion Criteria:

* Any autonomic cardiovascular, metabolic, neurologic, endocrine, or respiratory disease, that, in the opinion of the investigator, would exclude them from participation.
* Previously diagnosed liver and/or kidney dysfunction, including, but not limited to, acute and/or chronic kidney disease, cirrhosis, hepatitis, and fatty liver disease.
* Women who are pregnant or breastfeeding.
* Current use of tobacco or electronic cigarette, or regular (i.e., more than twice a week) use within the last 1 year.
* History of peripheral cold injury, skin disorder (eczema, psoriasis), or excessive tattooing.
* Known chronic (i.e., cancer, surgery) or acute conditions (i.e., diarrhea, constipation) of the rectum.
* Menthol allergy (described in detail in Section 7.0 and 9.0). Menthol can cause skin irritation when applied topically, especially for people with sensitive skin or allergies. For this reason, recruited participants will be screened for a menthol allergy during the informed consent/screening visit. We will apply a small quantity of the cream (~2ml) to an isolated body area to limit skin exposure. In the case a rash develops during the application of the cream, research staff will irrigate the area to remove the substance and limit further exposure. A 24-hour follow-up phone call initiated by research staff will be implemented to follow-up on all adverse reactions. Detectable BAT activation during a localized cold stress test (i.e., face cooling test) (procedure described in detail in Section 7.0).
* Using medications with direct effects on the cardiovascular system including, but not limited to:

  * Anticoagulants.
  * Antiplatelet agents.
  * ACE Inhibitors.
  * Angiotensin II receptor blockers.
  * Angiotensin-receptor neprilysin inhibitors.
  * Beta blockers.
  * Calcium, potassium, or sodium channel blockers.
  * Cholesterol lowering medications.
  * Digitalis preparations.
  * Diuretics.
  * Vasodilators.
  * Anticholinergics.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Resting energy expenditure | from prior to the interventions to 1 hour and 2 hours post gel application
  kcal/min
Infrared thermography supraclavicular skin temperature | from prior to the interventions to 1 hour and 2 hours post gel application
  temperature in degrees C
Shivering via electromyography | from prior to the interventions to 1 hour and 2 hours post gel application
  a percent of maximal activity

SECONDARY OUTCOMES:
Body temperatures | from prior to the interventions to 1 hour and 2 hours post gel application
  Combined intestinal and skin temperatures in degrees C
Skin blood flow | from prior to the interventions to 1 hour and 2 hours post gel application
  red blood cell flux
Cardiovascular measurements | from prior to the interventions to 1 hour and 2 hours post gel application
  heart rate in beats/min and blood pressure in millimeters of mercury
Thermal perceptions | from prior to the interventions to 1 hour and 2 hours post gel application
  assessed using Likert Scales thermal discomfort (1=comfortable; 4=very uncomfortable) and thermal sensation (1=cold; 4=neutral; 7=hot)

CONTACTS AND LOCATIONS:
Overall Officials: Blair D Johnson, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF